CLINICAL TRIAL: NCT01587677
Title: Diagnostic Evaluation of a Urine and Plasma Based LAM FLISA for the Diagnosis of Infection With Mycobacterium Tuberculosis
Brief Title: Evaluation of a LAM FLISA for the Diagnosis of Tuberculosis
Acronym: LAM FLISA
Status: Completed | Type: Observational
Sponsor: Research Center Borstel (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Principal Investigator, Christian Herzmann, Head of Clinical Trials Unit, Research Center Borstel
Other Study IDs: RCBorstel001
Record Dates: First submitted 2012-04-23; First posted 2012-04-30 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Tuberculosis
Keywords: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and EDTA plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Confirmed tuberculosis
- Confirmed non-tuberculous mycobacterial infection
- Confirmed bronchial carcinoma
- Suspected tuberculosis but confirmed alternative diagnosis

SUMMARY:
Tuberculosis is a bacterial infection causing 1.1 million deaths annually worldwide. Diagnosis of the disease is often time consuming or challenging. Many cases of tuberculosis require advanced and expensive diagnostic methods that restrict their availability in resource limited countries where the burden of tuberculosis is highest. The development of rapid point of care diagnostics is required.

Lipoarabinomannan (LAM) is part of the bacterial cell wall in M. tuberculosis. It is released when bacteria are multiplying or dying. LAM can be detected in the urine since it is filtered from the blood in the kidneys. The detection of LAM in the urine by conventional enzyme linked immuno-sorbent assay (ELISA) techniques was hampered in the past by a low sensitivity and multiple processing steps. Recently, fluorescence linked immuno-sorbent assay (FLISA) has been shown to detect LAM in concentrations that are several magnitudes lower that with ELISA based methods. Furthermore the procedure requires less separate steps for processing the sample.

This study aims to validate the new diagnostic test by comparing patients with (a) confirmed tuberculosis (n=25), (b) infection with non-tuberculous mycobacteria (n=25), (c) bronchial carcinoma (n=25), (d) suspected tuberculosis but confirmed alternative diagnosis (estimated n=20). Single blood and urine samples of these groups will be used to evaluate the sensitivity and specificity of the test.

In patients with confirmed tuberculosis the LAM FLISA will also be assessed as a biomarker for the monitoring of tuberculosis treatment success. Initially, 2-5 samples blood and urine are required during the first week, followed by twice weekly and weekly sampling intervals over a period of 12 weeks maximum. The study participation ends when the patient is discharged from hospital.

As a substudy, the blood samples will be used to evaluate an enzyme linked immuno-sorbent assay (ELISA) for the detection of lipid antigens that are specific for Mycobacterium tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected or confirmed infection with M. tuberculosis (MTB) or confirmed infection with non-tuberculous mycobacteria (NTM) or confirmed bronchial carcinoma
2. Oral and written consent to study participation (children: parent's consent)

Exclusion Criteria:

1. Inability to follow the study requirements
2. Patient in custodianship or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed or suspected tuberculosis. Patients with NTM infection or bronchial carcinoma serve as control
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Rate of patients with false positive and false negative urine LAM detection | On admission to hospital

SECONDARY OUTCOMES:
Rate of patients with false negative and false positive blood LAM detection | On admission to hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center Borstel, Borstel, Germany